CLINICAL TRIAL: NCT01375894
Title: Body Movement Imitation and Perspective Perception Among Psychiatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHA-07-11
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Schizophrenia; Depression
MeSH Terms: conditions — Schizophrenia; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- depresive patients (Active Comparator): 30 patients suffering from depression
  Interventions: Device: imitation assessment using the 5-dt "data glove".
- Schizophrenia patients (Experimental): 30 Schizophrenia patients
  Interventions: Device: imitation assessment using the 5-dt "data glove".

INTERVENTIONS:
Device: imitation assessment using the 5-dt "data glove". — measuring the speed of the hand during imitation

SUMMARY:
The ability to understand the other's perspective and respond accordingly is the most important normal process of daily social life and is probably one of the foundations of human existence. This capability is reflected, inter alia, as an imitation - an important and effective form of learning which is very developed in humans. When we are required to imitate a particular movement, speed of response depends on the perspective of the movement. Imitative response is implemented faster when the movement is observed from first-person perspective, than if the motion is presented from the perspective of a third party.

While healthy individuals don't find it difficult to imitate, or to understand the other's emotion expression, there are psychiatric populations (such as autism and schizophrenia) who find it difficult to demonstrate these capabilities (Park, Matthews et al. 2008). Beyond these capabilities impairment, schizophrenic patients have difficulty distinguishing between their arm movements and those of a foreign hand and find it difficult to leave the boundaries of egocentric interpretation of reality and adopt the other's point of view. These behavioral disorders arise from defects in the network of mirror neurons (Buccino and Amore 2008; Langdon, Coltheart et al. 2010).

Therefore, the investigator expect that schizophrenic patients will not see a preference for movements that will be displayed in first-person perspective from the same movements that will be displayed from the perspective of a third party. Consequently, the investigator speculate that these subjects will not exhibit differences at imitating the response of which will be presented from different perspectives (Jackson, Meltzoff et (al. 2006.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 20-65.
2. Subjects who met the criteria for diagnosis of major DSM-IV for schizophrenia or unipolar depression.
3. Subjects with normal or corrected vision.
4. Subjects who sign informed consent for their participation in the experiment

Exclusion Criteria:

1. Patients with acute disorder, or an unstable patient. Especially neurological disorders or head injuries.
2. Drug Abuse in the past year.
3. Lack of jurisdiction, such as people with mental retardation or dementia.
4. assessed with high suicide risk.
5. patients which are Compulsory hospitalized.
6. Pregnant women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
speed of hand movement according to the reaction glove | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel